CLINICAL TRIAL: NCT01090505
Title: Phase 2 Study of S-1 and Oxaliplatin as Neoadjuvant Chemotherapy for Locally Advanced
Brief Title: Study of S-1 and Oxaliplatin as Neoadjuvant Chemotherapy for Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: L Chen, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-ChinaPLAGH-2010
Record Dates: First submitted 2010-03-16; First posted 2010-03-22 (Estimated); Last update posted 2010-03-22 (Estimated); Status verified 2009-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug:S-1:80mg/m2;oxaliplatin 130mg/m2 (Experimental): Drug: Neoadjuvant chemotherapy(S-1+Oxaliplatin) followed by D2 gastrectomy
  Interventions: Drug: Drug: S-1 and oxaliplatin
- surgery (No Intervention): Procedure/Surgery: Gastrectomy with D2 dissection
  Interventions: Drug: Drug: S-1 and oxaliplatin

INTERVENTIONS:
Drug: Drug: S-1 and oxaliplatin — Drug:S-1:80mg/m2;oxaliplatin 130mg/m2
  Other Names: S-1:Taiho; Oxaliplatin：sanofi-aventis

SUMMARY:
The purpose of this study is to determine whether S-1 and oxaliplatin as neoadjuvant chemotherapy may improve survival benefit compared with control.

ELIGIBILITY:
Inclusion Criteria:

1. DISEASE CHARACTERISTICS:

   Histologically confirmed gastric adenocarcinoma Locally advanced disease:Clinical stage T3-4, N0-3, M0 (according to the Japanese gastric cancer classification)
2. Planning to undergo gastric cancer D2 surgery after neoadjuvant chemotherapy
3. Age:20 to 75
4. Performance status:ECOG 0-2
5. Life expectancy:Not specified
6. Hematopoietic:WBC 4,000-12,000/mm^3；Granulocyte count ≥ 2,000/mm^3；Platelet count ≥ 100,000/mm^3；Hemoglobin ≥ 9.0 g/dL;Hepatic:AST and ALT ≤ 100 U/L；Bilirubin ≤ 1.5 mg/dL
7. Adequate organ function
8. Able to swallow oral medication
9. Written informed consent

Exclusion Criteria:

1. Synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ
2. Pregnant or breast-feeding women
3. Severe mental disease
4. Systemic administration of corticosteroids, flucytosine, phenytoin or warfarin
5. Other severe complications such as paralytic ileus, intestinal pneumonitis, pulmonary fibrosis, or ischemic heart disease
6. Myocardial infarction within six disease-free months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years

SECONDARY OUTCOMES:
response rate | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- China PLA General Hospital, Beijing, Beijing Municipality, China